CLINICAL TRIAL: NCT00920348
Title: The Canadian Cohort Obstructive Lung Disease
Acronym: CanCOLD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); GlaxoSmithKline (Industry); AstraZeneca (Industry); Pfizer (Industry); Boehringer Ingelheim (Industry); Novartis (Industry); Takeda (Industry); Merck Sharp & Dohme LLC (Industry); Almirall, SAS (Industry)
Responsible Party: Principal Investigator, Jean Bourbeau, MD, M.Sc., McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: IRO-93326
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: COPD; Chronic Obstructive Pulmonary Disease
Keywords: Chronic obstructive pulmonary disease; COPD; Cohort study; prospective longitudinal study; tissue bank
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sampling
  * Biomarkers:IL-6, CRP, CC-16, SP-D"
  * DNA for genetics, epigenetic and RNA for transcriptomics
  * Markers for cardiovascular diseases: LDL, LDL and HDL sizes, Apo B, Apo A1, CRP, IL6, TNF alpha, Adiponectine, Leptine, Glucose and Insulin.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Group 1: COPD moderate-severe(GOLD2-4)(post-BD FEV1/FVC<0.70 and FEV1<80% of pred.)
- Group 2: COPD mild (GOLD1)(post-BD FEV1/FVC<0.70 AND FEV1>=80% of pred.)
- Group 3: COPD at risk (ever smoker with post-BD FEV1/FVC>=0.70)
- Group 4: "Healthy control" never smokers without respiratory disease (post-BD FEV1/FVC>=0.70.

SUMMARY:
Abstract Chronic obstructive pulmonary disease (COPD) is the fourth leading cause of death in Canada. COPD is not just a disease of men, nor is it solely a disease in old age. Women have been underrepresented and early disease has not been studied. Underdiagnosis of COPD remains a significant problem, and it may indicate an unmet healthcare need. This can potentially results not only in a patient been misinformed, but can lead to incorrect management.

Epidemiological research is needed to develop a framework to combat this major health problem, by better characterization of the population of men and women at risk and patients with early disease, by better understanding which factors modifiable through health interventions are related to health perception (health-related quality of life) and disease evolution.

This will be possible through a nationwide study, the Canadian Cohort Obstructive Lung disease (CanCOLD), a prospective longitudinal study. The CanCOLD study is built on the current ongoing prevalence nationwide study, the Canadian Obstructive Lung disease "COLD" study.

The CanCOLD will be the first study to assess prevalence of disease across Canada and its consequence in men and women, and to evaluate a conceptual model of disease severity based on patient's health perception (health-related quality of life). Ultimately, this project will extend to a longitudinal follow up (3 years or beyond) and will allow to have a better understanding of the lifestyle risk factors, not only smoking but also diet, physical activity, and co morbid conditions. This will be a great asset to shift from management of a single risk factor (tobacco control) to total COPD risk management. The results of the study will greatly help to assist decision makers in developing policies to improve the diagnosis, the management of COPD and to optimize health care services use.

ELIGIBILITY:
Inclusion Criteria:

* All the subjects have taken part in the COLD study, a true population based prevalence study. Subjects must have an inclusion criteria of 40 years and older to participate in the COLD study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects' selection and participation in CanCOLD- longitudinal cohort: Subjects will be recruited from the study site participants (total from cross-sectional ≈5,000 subjects, men and women).
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2010-01; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
What risk factors other than smoking determine the development and progression of COPD. | One visit a year every 18 months

SECONDARY OUTCOMES:
What are the combinations of the disease and patient attributes that differentiate individuals (men/women) with COPD as they relate to relevant outcomes (symptoms, exacerbations, disease progression or death) | One visit a year 18 months
Is early detection of COPD with spirometry meaningful according to sex and ageing. | One visit a year 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean Bourbeau, M.D., M.Sc., Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Wan Tan, M.D., Principal Investigator — CAAA University of British Columbia; François Maltais, M.D., Principal Investigator — CFBA Université Laval; Shawn Aaron, M.D., M.Sc., Principal Investigator — OHGC Ottawa Hospital General Campus; Denis O'Donnell, M.D., Principal Investigator — CEDA Queen's University (Kinsgston); Darcy D Marciniuk, M.D., Principal Investigator — CCAA University of Saskatchewan; Robert Cowie, M.D., Principal Investigator — CBBA University of Calgary; Kenneth R. Chapman, M.D., M.Sc., Principal Investigator — CEAA University of Toronto; Paul Hernandez, M.D., Principal Investigator — CHAA Dalhousie University (Nova Scotia); Mark J. FitzGerald, M.D., Principal Investigator — CAAA University of British Columbia; Donald Sin, M.D., Principal Investigator — CAAA University of British Columbia; Andrea Benedetti, Ph.D., Principal Investigator — INUD McGill University Healty Center; Yves Lacasse, M.D., M.Sc., Principal Investigator — CPVR Institut universitaire de cardiologie et de pneumologie de Québec; Pierre Ernst, M.D., Principal Investigator — McGill University; Harvey Coxson, M.D., Principal Investigator — University of British Columbia; Roger Goldstein, M.D., Principal Investigator — CEAA University of Toronto; Carlo Marra, Ph.D., Principal Investigator — CAAA University of British Columbia
Locations (9):
- Canada (9):
  - Health Sciences Centre, Calgary, Alberta
  - St-Paul's Hospital, Vancouver, British Columbia
  - Halifax Infirmary, Halifax, Nova Scotia
  - Kingston General Hospital, Kingston, Ontario
  - Ottawa Hospital General, Ottawa, Ontario
  - University of Toronto, Toronto, Ontario
  - Montreal Chest Institute, Montreal, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
  - Institut universitaire de cardiologie et de pneumologie de Québec, Québec

IPD SHARING:
Plan to Share IPD: Yes
publications; data sharing through substudies submission

REFERENCES:
- [Derived] Cordero AIH, Li X, Yang CX, Ambalavanan A, MacIsaac JL, Kobor MS, Doiron D, Tan W, Bourbeau J, Sin DD, Duan Q, Leung JM; CanCOLD Collaborative Research Group. Cannabis smoking is associated with persistent epigenome-wide disruptions despite smoking cessation. BMC Pulm Med. 2025 Apr 9;25(1):168. doi: 10.1186/s12890-025-03634-9. PMID 40205553
- [Derived] Ekstrom M, Lewthwaite H, Li PZ, Bourbeau J, Tan WC, Jensen D; CanCOLD Collaborative Research Group. Identifying Abnormal Exertional Breathlessness in COPD: Comparing Modified Medical Research Council and COPD Assessment Test With Cardiopulmonary Exercise Testing. Chest. 2025 Mar;167(3):697-711. doi: 10.1016/j.chest.2024.10.027. Epub 2024 Oct 28. PMID 39490971
- [Derived] Virdee S, Tan WC, Hogg JC, Bourbeau J, Hague CJ, Kirby M; CanCOLD Collaborative Research Group. CT Chest Imaging Using Normalized Join-Count: Predicting Emphysema Progression in the CanCOLD Study. Radiology. 2024 Jul;312(1):e233265. doi: 10.1148/radiol.233265. PMID 39012250
- [Derived] Phillips DB, James MD, Vincent SG, Elbehairy AF, Neder JA, Kirby M, Ora J, Day AG, Tan WC, Bourbeau J, O'Donnell DE; CanCOLD Collaborative Research Group and the Canadian Respiratory Research Network. Physiological Characterization of Preserved Ratio Impaired Spirometry in the CanCOLD Study: Implications for Exertional Dyspnea and Exercise Intolerance. Am J Respir Crit Care Med. 2024 Jun 1;209(11):1314-1327. doi: 10.1164/rccm.202307-1184OC. PMID 38170674
- [Derived] Abozid H, Kirby M, Nasir N, Hartl S, Breyer-Kohansal R, Breyer MK, Burghuber OC, Bourbeau J, Wouters EFM, Tan W; CanCOLD Collaborative research Group and the Canadian Respiratory Research Network. CT airway remodelling and chronic cough. BMJ Open Respir Res. 2023 May;10(1):e001462. doi: 10.1136/bmjresp-2022-001462. PMID 37173074
- [Derived] Ross BA, Doiron D, Benedetti A, Aaron SD, Chapman K, Hernandez P, Maltais F, Marciniuk D, O'Donnell DE, Sin DD, Walker BL, Tan W, Bourbeau J; CanCOLD Collaborative Research Group and the Canadian Respiratory Research Network. Short-term air pollution exposure and exacerbation events in mild to moderate COPD: a case-crossover study within the CanCOLD cohort. Thorax. 2023 Oct;78(10):974-982. doi: 10.1136/thorax-2022-219619. Epub 2023 May 5. PMID 37147124
- [Derived] Krishnan S, Tan WC, Farias R, Aaron SD, Benedetti A, Chapman KR, Hernandez P, Maltais F, Marciniuk DD, O'Donnell DE, Sin DD, Walker B, Bourbeau J; Canadian Cohort Obstructive Lung Disease Collaborative Research Group and the Canadian Respiratory Research Network. Impaired Spirometry and COPD Increase the Risk of Cardiovascular Disease: A Canadian Cohort Study. Chest. 2023 Sep;164(3):637-649. doi: 10.1016/j.chest.2023.02.045. Epub 2023 Mar 4. PMID 36871842
- [Derived] Moslemi A, Makimoto K, Tan WC, Bourbeau J, Hogg JC, Coxson HO, Kirby M; Canadian Cohort of Obstructive Lung Disease. Quantitative CT Lung Imaging and Machine Learning Improves Prediction of Emergency Room Visits and Hospitalizations in COPD. Acad Radiol. 2023 Apr;30(4):707-716. doi: 10.1016/j.acra.2022.05.009. Epub 2022 Jun 8. PMID 35690537
- [Derived] Phillips DB, Elbehairy AF, James MD, Vincent SG, Milne KM, de-Torres JP, Neder JA, Kirby M, Jensen D, Stickland MK, Guenette JA, Smith BM, Aaron SD, Tan WC, Bourbeau J, O'Donnell DE; CanCOLD Collaborative Research Group and the Canadian Respiratory Research Network. Impaired Ventilatory Efficiency, Dyspnea, and Exercise Intolerance in Chronic Obstructive Pulmonary Disease: Results from the CanCOLD Study. Am J Respir Crit Care Med. 2022 Jun 15;205(12):1391-1402. doi: 10.1164/rccm.202109-2171OC. PMID 35333135
- [Derived] Tan WC, Bourbeau J, Nadeau G, Wang W, Barnes N, Landis SH, Kirby M, Hogg JC, Sin DD; CanCOLD Collaborative Research Group; authors would also like to thank the men and women who participated in the study and individuals in the CanCOLD Collaborative Research Group not listed as authors:. High eosinophil counts predict decline in FEV1: results from the CanCOLD study. Eur Respir J. 2021 May 27;57(5):2000838. doi: 10.1183/13993003.00838-2020. Print 2021 May. PMID 33303555
- [Derived] Lewthwaite H, Elsewify O, Niro F, Bourbeau J, Guenette JA, Maltais F, Marciniuk DD, O'Donnell DE, Smith BM, Stickland MK, Tan WC, Jensen D; CanCOLD Collaborative Research Group; Canadian Respiratory Research Network. Normative Cardiopulmonary Exercise Test Responses at the Ventilatory Threshold in Canadian Adults 40 to 80 Years of Age. Chest. 2021 May;159(5):1922-1933. doi: 10.1016/j.chest.2020.11.009. Epub 2020 Nov 18. PMID 33217419
- [Derived] Barrecheguren M, Pinto L, Mostafavi-Pour-Manshadi SM, Tan WC, Li PZ, Aaron SD, Benedetti A, Chapman KR, Walker B, Fitzgerald JM, Hernandez P, Maltais F, Marciniuk DD, O'Donnell DE, Sin DD, Bourbeau J; CanCOLD Collaborative Research Group and the Canadian Respiratory Research Network. Identification and definition of asthma-COPD overlap: The CanCOLD study. Respirology. 2020 Aug;25(8):836-849. doi: 10.1111/resp.13780. Epub 2020 Feb 16. PMID 32064708
- [Derived] Gupta N, Pinto L, Benedetti A, Li PZ, Tan WC, Aaron SD, Chapman KR, FitzGerald JM, Hernandez P, Marciniuk DD, Maltais F, O'Donnell DE, Sin D, Walker BL, Bourbeau J; Canadian Respiratory Research Network and the CanCOLD Collaborative Research Group. The COPD Assessment Test: Can It Discriminate Across COPD Subpopulations? Chest. 2016 Nov;150(5):1069-1079. doi: 10.1016/j.chest.2016.06.016. Epub 2016 Jun 27. PMID 27364603
- [Derived] Tan WC, Sin DD, Bourbeau J, Hernandez P, Chapman KR, Cowie R, FitzGerald JM, Marciniuk DD, Maltais F, Buist AS, Road J, Hogg JC, Kirby M, Coxson H, Hague C, Leipsic J, O'Donnell DE, Aaron SD; CanCOLD Collaborative Research Group. Characteristics of COPD in never-smokers and ever-smokers in the general population: results from the CanCOLD study. Thorax. 2015 Sep;70(9):822-9. doi: 10.1136/thoraxjnl-2015-206938. Epub 2015 Jun 5. PMID 26048404